CLINICAL TRIAL: NCT03892213
Title: A Phase 1 Pharmacokinetic Drug-Drug Interaction Study of Benznidazole and E1224 in Healthy Male Volunteers
Brief Title: Pharmacokinetic Drug-Drug Interaction Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: PhinC Development (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNDi-CH-E1224-002
Record Dates: First submitted 2014-08-20; First posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Chagas Disease
Keywords: Chagas Disease; drug-drug interaction; benznidazole; E1224; pharmacokinetics
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Benznidazole and E1224 (Other): Benznidazole and E1224
  Interventions: Drug: Benznidazole; Drug: E1224

INTERVENTIONS:
Drug: Benznidazole — Benznidazole single dose (2.5 mg/kg) at Day 1. Benznidazole single dose (2.5 mg/kg) at Day 9*. Benznidazole multiple dose (2.5 mg/kg twice daily) from Day 12* until Day 15.
  Other Names: Abarax® (Benznidazole 100mg or 50mg).
Drug: E1224 — E1224 multiple dose 400 mg loading dose once daily for 3 days (i.e. from Day 4 to Day 6 followed by maintenance dose 100mg once daily for 9 days (from Day 7 to Day15).
  On Day 9 and from Day 12 to Day 15, E1224 and benznidazole will be given concomitantly.
  Other Names: E1224 is a prodrug monolysine form of ravuconazole.

SUMMARY:
The purpose of this study is to determine whether benznidazole and E1224 should be administered concomitantly in patients with Chagas Disease as not enough data are available. This study aims to assess cross interactions of these two compounds.

DETAILED DESCRIPTION:
Benznidazole and E1224 are intended to be administered concomitantly in patients with Chagas disease. Thus, an in vivo interaction study in healthy volunteers may be justified as the two drugs are intended to be administered concomitantly in patients and no in vivo nor in vitro data are available.

In addition both interactions (potential for benznidazole to interact on the pharmacokinetic (PK) of E1224 and potential for E1224 on the PK of benznidazole should be studied.

Benznidazole t1/2 is quite short (12 h) whereas E1224 t1/2 is very long (more than 200 h). Therefore it was chosen to study the interaction of E1224 at steady-state while interaction of benznidazole after single dose appears more appropriate instead of a classical randomized cross-over design.

ELIGIBILITY:
Inclusion Criteria:

1. Male healthy volunteers 18 to 45 years of age;
2. Light smokers (less than 5 cigarettes per day) or subjects who are non-smokers;
3. Male subjects with a body weight of at least 50 kg and a body mass index (BMI) calculated as weight in kg/height (in m2) from 18 to 28 kg/m2 at screening;
4. Able to communicate well with the Investigator and research staff and to comply with the requirements of the entire study;
5. Provision of written informed consent to participate as shown by a signature on the volunteer consent form;

Exclusion Criteria:

1. Who on direct questioning and physical examination have evidence of any clinically significant acute or chronic disease, including known or suspected HIV, hepatites B virus (HBV) or hepatites C virus (HCV) infection;
2. Who has positive diagnosis of T. cruzi infection indicated by Conventional serology;
3. With any clinically significant abnormality following review of pre-study laboratory tests, vital signs, full physical examination and 12-lead ECG;
4. Who forfeit their freedom by administrative or legal award or who were under guardianship;
5. Unwilling to give their informed consent;
6. Who have a positive laboratory test for Hepatitis B surface antigen (HbsAg), or anti-HIV 1/2 or anti- HCV antibodies;
7. Who have a history of allergy (serious or not), allergic skin rash, asthma, intolerance, sensitivity or photosensitivity to any drug;
8. Who are known or suspected alcohol or drug abusers (more than 14 units of alcohol per week, one unit = 8 g or about 10 mL of pure alcohol);

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration (Cmax) of Benznidazole | Day 1 and day 9
  BNZ PK parameter following single dose to investigate the possible drug-drug interaction between BNZ and E1224 through evaluation of the PK characteristics of both drugs when given alone or concomitantly.
Time of occurrence of maximum plasma concentration (tmax) of Benznidazole | Day 1 and day 9
  BNZ PK parameter following single dose to investigate the possible drug-drug interaction between BNZ and E1224 through evaluation of the PK characteristics of both drugs when given alone or concomitantly.
Area under the serum concentration versus time curve from time zero to the time (t) corresponding to the last quantifiable concentration (AUC 0-t) of Benznidazole | Day 1 and day 9
  BNZ PK parameter following single dose to investigate the possible drug-drug interaction between BNZ and E1224 through evaluation of the PK characteristics of both drugs when given alone or concomitantly.
Area under the concentration-time curve from time zero to infinity with extrapolation of the terminal phase (AUC 0-∞) of Benznidazole | Day 1 and day 9
  BNZ PK parameter following single dose to investigate the possible drug-drug interaction between BNZ and E1224 through evaluation of the PK characteristics of both drugs when given alone or concomitantly.
Terminal half-life (t1/2) of Benznidazole | Day 1 and day 9
  BNZ PK parameter following single dose to investigate the possible drug-drug interaction between BNZ and E1224 through evaluation of the PK characteristics of both drugs when given alone or concomitantly.
Maximum serum concentration (Cmax) of Ravuconazole. | Day 8 and day 15, day 6 (morning pre-dose), day 7 (morning pre-dose), day 8 (morning pre-dose), day 13 (morning pre-dose), day 14 (morning pre-dose), and day 15 (morning pre-dose)
  PK parameter of ravuconazole following multiple dose to investigate the possible drug-drug interaction between BNZ and E1224 (prodrug of ravuconazole) through evaluation of the PK characteristics of both drugs when given alone or concomitantly.
Time of occurrence of maximum plasma concentration (tmax) of Ravuconazole. | Day 8 and day 15, day 6 (morning pre-dose), day 7 (morning pre-dose), day 8 (morning pre-dose), day 13 (morning pre-dose), day 14 (morning pre-dose), and day 15 (morning pre-dose)
  PK parameter of ravuconazole following multiple dose to investigate the possible drug-drug interaction between BNZ and E1224 (prodrug of ravuconazole) through evaluation of the PK characteristics of both drugs when given alone or concomitantly.
The area under the blood drug concentration vs. time curve from time zero (pre-dose) to 24 h post-dose (AUC 0-24) | Day 8 and day 15, day 6 (morning pre-dose), day 7 (morning pre-dose), day 8 (morning pre-dose), day 13 (morning pre-dose), day 14 (morning pre-dose), and day 15 (morning pre-dose)
  PK parameter of ravuconazole following multiple dose to investigate the possible drug-drug interaction between BNZ and E1224 (prodrug of ravuconazole) through evaluation of the PK characteristics of both drugs when given alone or concomitantly.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Through study completion, i.e up to 22 days.
  Monitoring for the occurrence of adverse events (AEs)
Clinically significant alterations in pulse rate | Through study completion, i.e up to 22 days.
  Parameter to assess the safety and tolerability of multiple oral doses of BNZ and E1224 given in healthy male subjects.
Clinically significant alterations in blood pressure | Through study completion, i.e up to 22 days.
  Parameter to assess the safety and tolerability of multiple oral doses of BNZ and E1224 given in healthy male subjects.
Clinically significant alterations in 12-lead ECG | Through study completion, i.e up to 22 days.
  Parameter to assess the safety and tolerability of multiple oral doses of BNZ and E1224 given in healthy male subjects
Clinically significant Haematology abnormalities (hemoglobin, RBC, hematocrit, MCV, MCH, MCHC, WBC, including differential, platelet counts) | Day 1, Day 4, Day 7, Day 9, Day 10, Day 12, Day 13, Day 14 and Day 15 pre morning dose
  Parameter to assess the safety and tolerability of multiple oral doses of BNZ and E1224 given in healthy male subjects.
Clinically significant Biochemistry abnormalities (albumin (ALB), ALP, ALT, AST, gamma-glutamyl transferase (GGT), chlorides (Cl-), creatinine, glucose (GLU), potassium (K+), sodium (Na+), total bilirubin (TBIL), total proteins (TP), Urea. | Day 1, Day 4, Day 7, Day 9, Day 10, Day 12, Day 13, Day 14 and Day 15 pre morning dose
  Parameter to assess the safety and tolerability of multiple oral doses of BNZ and E1224 given in healthy male subjects.
Clinically significant Urinalysis abnormalities (leukocytes, pH, proteins, urobilinogen, blood, nitrites, glucose, ketone bodies, bilirubin). | Screening and day 22
  Parameter to assess the safety and tolerability of multiple oral doses of BNZ and E1224 given in healthy male subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Isabela Ribeiro, MD, Study Chair — Drugs for Neglected Diseases initiative; Ethel Feleder, MD, Principal Investigator — F.P. Clinical Pharma Clinical Research Unit
Locations (1):
- FP Clinical Pharma - Juncal 4484 - 3o piso, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided